CLINICAL TRIAL: NCT02258035
Title: Isolation of Genotype-specific Isoforms of Human Vitamin D-binding Protein (DBP/Gc)
Brief Title: Isolation of Vitamin D Binding Protein Isoforms From Human Volunteers
Status: Active, not recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s57027
Record Dates: First submitted 2014-09-26; First posted 2014-10-07 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D binding protein (DBP)
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum will be derived from 100-150 ml of blood and used for protein purification
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- DBP/Gc1f-1f genotype: Human volunteers homozygous for the 1f-1f (fast) genotype of DBP.
  Interventions: Other: Blood draw
- DBP/Gc1s-1s genotype: Human volunteers homozygous for the 1s-1s (slow) genotype of DBP.
  Interventions: Other: Blood draw
- DBP/Gc 2-2 genotype: Human volunteers homozygous for the 2-2 genotype of DBP.
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — Sampling of 100-150 ml of blood

SUMMARY:
The purpose of this study is to isolate genotype-specific DBP/Gc from homozygous human volunteers and use these purified proteins to cross-validate existing or novel assays for this serum protein and to evaluate the binding characteristics of these variants of DBP/Gc for different vitamin D metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy adults (≥ 18 years), non pregnant, with known DBP/Gc genotype

Exclusion Criteria:

* Inability to provide written informed consent
* No children or pregnant women
* Persons with known abnormal serum proteins

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with known genotype of DBP/Gc, as identified in the clinical database of the Multidisciplinary Breast Centre, University Hospitals Leuven, and free of breast cancer recurrence at the time of blood sampling.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Vitamin D binding protein binding characteristics (affinity constant) | single blood draw at time of consultation, an expected average 4 years after curative treatment for breast cancer
  In vitro characterization

SECONDARY OUTCOMES:
Correlation coefficient (r) of different DBP assays | single blood draw at time of consultation, an expected average 4 years after curative treatment for breast cancer
  In vitro characterization

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Vanderschueren, MD PhD, Principal Investigator — UZ Leuven; Roger Bouillon, MD PhD, Study Chair — UZ Leuven; Hans Wildiers, MD PhD, Study Chair — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

REFERENCES:
- [Background] Hatse S, Lambrechts D, Verstuyf A, Smeets A, Brouwers B, Vandorpe T, Brouckaert O, Peuteman G, Laenen A, Verlinden L, Kriebitzsch C, Dieudonne AS, Paridaens R, Neven P, Christiaens MR, Bouillon R, Wildiers H. Vitamin D status at breast cancer diagnosis: correlation with tumor characteristics, disease outcome, and genetic determinants of vitamin D insufficiency. Carcinogenesis. 2012 Jul;33(7):1319-26. doi: 10.1093/carcin/bgs187. Epub 2012 May 23. PMID 22623648